CLINICAL TRIAL: NCT05679947
Title: The Effect of Mobilization Protocol Developed for Knee Arthroplasty Patients on Nursing Care-Sensitive Patient Outcomes
Brief Title: Mobilization Protocol for Knee Arthroplasty Patients
Acronym: KA-Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Bozok University (Other)
Responsible Party: Principal Investigator, Sevil Güler, Assoc. Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-77082166-604.01.02-140038
Record Dates: First submitted 2022-12-18; First posted 2023-01-11 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pain; Anxiety; Physical Function; Mobility; Arthroplasty
Keywords: knee arthroplasty; nursing; mobilization protocol; patient outcome; nurse sensitive outcomes; orthopaedic and trauma nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, parallel group single blinded, randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: the researcher learned the study and control groups after the pre-test data. The study group was trained with the mobilization protocol. The control group received training on the current mobilization procedure of the clinic. Participants did not know which group they were in.
  Outcomes Assessor. Study and control groups data were coded into the SPSS programme as group one and group two. Analysis of data was done by an independent statistician. The statistician has no information about which group the patients belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Protocol (Experimental): The study group patients were mobilized according to the developed mobilization protocol.The protocol includes six levels. Protocol levels are applied from the day the patient is operated and ends on the discharged day. The researcher explains the protocol levels to the patient before surgery.The patient is mobilized within the first 24 h after surgery. Implement mobilization protocol 3 times during the day and more as tolerated. Mobilization protocol:Level 1: Repositioning should occur every 2 h. Level 2: ROM should occur at least 3 times a day. Level 3: The head of bed (HOB) >30 degrees. Duration goal: 5-15 min. HOB 65≥ degrees with patient sit in the bed. Duration goal: 5-15 min. Progress to level 4. Level 4: HOB 65≥ degrees with legs in dependent position (recliner chair). Duration goal: 5-15 min. Progress to level 5. Level 5: Stand/pivot/step to chair. Sitting in chair. Duration goal: 5-15 min. Progress to level 6. Level 6: Patient is able to ambulate at least 3 times a day.
  Interventions: Other: Mobilization protocol
- Control (No Intervention): No intervention was made to the control group, only data were collected at the same time as the study group.The patients in the control group was mobilized by the researchers according to the routine clinical mobilization practice.

INTERVENTIONS:
Other: Mobilization protocol — The mobilization protocol includes six levels. Protocol levels are applied from the day the patient is operated and ends on the day of discharge. The researcher explains the protocol levels to the patient before surgery.The patient is mobilized within the first 24 hours after surgery. Implement mobilization protocol three times during the day and more as tolerated. Mobilization protocol:Level 1: Repositioning should occur every two hours. Level 2: Range of motion (PROM) should occur at least three times a day. Level 3: The head of bed (HOB) >30 degrees. Duration goal: 5-15 minutes. HOB 65≥ degrees with patient sit in the bed. Duration goal: 5-15 minutes. Progress to level 4. Level 4: HOB 65≥ degrees with legs in dependent position (recliner chair). Duration goal: 5-15 minutes. Progress to level 5. Level 5: Stand/pivot/step to chair. Sitting in chair. Duration goal: 5-15 minutes. Progress to level 6. Level 6: Patient is able to ambulate at least three times a day.
  Arms: Mobilization Protocol

SUMMARY:
This randomized controlled study evaluates the effect of mobilization protocol applied to knee arthroplasty patients on anxiety level, pain, mobility and functional status.

DETAILED DESCRIPTION:
In the study, 68 knee arthroplasty patients were randomly assigned to the study and control groups. The mobilization protocol was applied to the study group (34). The mobilization protocol starts on the day of the operation and is completed on the day of discharge. The patient is mobilized within the first 24 hours after surgery. Mobilization protocol includes six levels. Level 1: Repositioning should occur every two hours. Level 2: Range of motion (PROM) should occur at least three times a day. Level 3: The head of bed (HOB) >30 degrees. Duration goal: 5-15 minutes. HOB 65≥ degrees with patient sit in the bed. Duration goal: 5-15 minutes. Progress to level 4. Level 4: HOB 65≥ degrees with legs in dependent position (recliner chair). Duration goal: 5-15 minutes. Progress to level 5. Level 5: Stand/pivot/step to chair. Sitting in chair. Duration goal: 5-15 minutes. Progress to level 6. Level 6: Patient is able to ambulate at least three times a day. No intervention was applied to the control group. The primary outcome of the study is the effect of mobilization protocol on the state anxiety level, pain, mobility and physical function of knee arthroplasty patients. The results collected before the mobilization protocol, postoperative first day, second day, the discharged day and the 3rd week after discharge.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to participate in research

Being 18 years or older

Having unilateral elective knee arthroplasty surgery

Having DA surgery for the first time

It is the absence of an obstacle to communicating cognitively, emotionally and verbally.

Exclusion Criteria:

Patients who initially agreed to participate in the study but wished to leave later were excluded from the study.

In the event of a complication affecting the mobilization of the patient during the intraoperative and post-operative period, the patient is excluded from the study.

He was excluded from the study due to the development of a cognitive, emotional and verbal barrier to communication after the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Inventory | Change State-Anxiety scale points at 3 weeks
  The State-Anxiety scale consists of twenty statements that evaluate how respondents' feel about anxiety "right now, at this moment" through four scales: one (not at all), two (somewhat), three (moderately so), and four (very much so). A rating of four indicates the presence of a high level anxiety and one indicates the absence of a high level anxiety. The anxiety level was found by calculation of scores, The range of scores is from 20-80, the higher the score indicating greater anxiety
Pain evaluated using the Vizüel Analog Scale (VAS) | Change Pain scale points at 3 weeks
  The patient marks his or her own pain on a 10 cm ruler with painlessness on one end and the most severe pain on the other.
Physical function evaluated using knee injury and osteoarthritis outcome score-physical function short-form (KOOS-PS) | Change KOOS-PS scale points at 3 weeks
  The KOOS-PS scale is used to evaluate the activities of daily living and physical function of people due to osteoarthritis and knee injuries. Patients reported the degree of difficulty they had experienced due to knee pain in the previous week: 1) getting out of bed, 2) wearing socks/pantyhose, 3) getting up from sitting position, 4) bending down, 5) bending/rotating the injured knee while on the injured knee, 6) knee sitting on top and 7) squatting. All items are scored on a 5-point Likert scale (none, mild, moderate, severe, extreme) between 0-4. Each question is scored between 0-4. The raw score is the sum of 7 items. The range score from 0-100 is obtained using a conversion table.
Patient Mobility Scale | Change Patient Mobility scale scores at 2 days
  The Patient Mobility Scale measures the pain and difficulty associated with four postoperative activities: (1) turning in bed, (2) sitting at the side of the bed, (3) standing, and (4) walking. by using separate 15-cm visual analog scales with word descriptors placed along the length of the scale.
Observer Mobility Scale | Change Observer Mobility scale scores at 2 days
  The Observer Mobility Scale rates the degree of independence to dependence with numbers from 1 to 5 during performance of the four postoperative activities: (1) turning in bed, (2) sitting at the side of the bed, (3) standing, and (4) walking. A rating of 1 means the patient performs the activity independently without verbal prompting or assistance, and the rating of 5 means the patient is unable to perform the activity regardless of assistance or verbal prompting. The rank scores for turning, sitting, standing, and walking are summed, and a mean score is calculated for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinç Meşe, MASTER, Principal Investigator — Yozgat Bozok Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Turkey, Yozgat Bozok University, Yozgat Cıty Hospıtal, Yozgat
  - Yozgat Bozok University, Yozgat Cıty Hospıtal, Yozgat

IPD SHARING:
Plan to Share IPD: No